CLINICAL TRIAL: NCT04130945
Title: Effect of Erector Spina Plane Block on Cost of Laparoscopic Cholesistectomy Anesthesia
Brief Title: Cost Effect of Erector Spina Plane Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kırıkkale University (Other)
Responsible Party: Principal Investigator, Kevser Peker, assitant professor, Kırıkkale University
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: cost effectiveness
Record Dates: First submitted 2019-10-16; First posted 2019-10-18 (Actual); Last update posted 2020-07-01 (Actual); Status verified 2020-06

CONDITIONS: Cost Effectiveness
MeSH Terms: interventions — Costs and Cost Analysis

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group 1 (Active Comparator): patients with erector spine plane block
  Interventions: Other: erector spina plane block, cost analysis
- group 2 (No Intervention): patients without erector spine plane block

INTERVENTIONS:
Other: erector spina plane block, cost analysis — in preopererative period, ESP block is going to utilise for postoperative analgesia for patients who undergo laparoscopic procedure and cost analysis will make after the end of 24 hour of operation
  Arms: group 1

SUMMARY:
Use of erector spina plane (ESP) block for postoperative analgesia is continuously increasing. However, few studies have investigated intraoperative effects of ESP block. The investigators aim to study the effects of ESP block in terms of cost-effectiveness, consumption of inhalation agents and opioids in perioperative and postoperative period.

DETAILED DESCRIPTION:
Erector spina plane (ESP) block has analgesic efficiency and its popularity is growing steadily. ESP block forms a sensorial block by local anesthetic infiltration between the musculus erector spina and facia. ESP block given to participants undergoing laparoscopic cholecystectomy for postoperative opioid analgesia resulted in a decrease of postoperative pain scores in the first 24 h. Due to increases in health expenditure, cost control is becoming more and more important. Cost-effective studies are important in healthcare economics. Inhaled anesthetics used in anesthesia departments account for about 20% of total anesthetic agents. Local anesthetic agents decrease the minimum alveolar concentration (MAC) value of inhaled agents. And also in perioperative and post operative period, the anesthetic management often need to be supported with opioid drugs. The investigators think that ESP block has analgesic effects and decreases the consumption of inhalation agents. The investigators aim to investigate the cost-effectiveness of ESP block in anesthetic applications in laparoscopic procedures.

ELIGIBILITY:
Inclusion Criteria:

1. American Society of Anesthesiologist (ASA) physical status I-II,
2. ages 18-75 years,
3. undergoing laparoscopic cholecystectomy

Exclusion Criteria:

1. Patients with cardiac, endocrinological, neurological diseases,
2. patients with coagulation disorders
3. allergy to local anesthetics
4. Operations that started as laparoscopy but transitioned to open surgery for a surgical reason

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2019-09-11 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2019-11-30 (Actual)

PRIMARY OUTCOMES:
the formula of consumption of inhaled agent | 30 minute after the operation
  the formula which includes fresh gas flow, valume of inhaled agent vapor, sevoflurane concentration

CONTACTS AND LOCATIONS:
Overall Officials: Kevser Peker, Principal Investigator — Kırıkkale University Faculty of Medicine
Locations (1):
- Kırıkkale Univercity Faculty of Medicine Hospital, Kırıkkale, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No